CLINICAL TRIAL: NCT06742060
Title: A Study on the Trend of Serum Copeptin Levels and Its Clinical Value for Postoperative Central Diabetes Insipidus in Pediatric Patients After Neurosurgical Intervention in Intensive Care Unit
Brief Title: The Trend of Copeptin Levels and Its Clinical Value for Postoperative CDI in Pediatric Patients After NSI in ICU
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-30
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Insipidus, Neurohypophyseal; Copeptin Blood Levels; Copeptin; Neurosurgical Intervention
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum copeptin levels — For children who met the entry criteria, the blood samples were collected preoperatively (T0), 1h postoperatively (T1), 1 day postoperatively (T2), 2 days postoperatively (T3), 3 days postoperatively (T4), 4 days postoperatively (T5), 5 days postoperatively (T6) to test serum and peptide levels.

SUMMARY:
Central diabetes insipidus (CDI),a disease caused by the decrease of AVP (a hormone involved in the control of water-electrolyte balance ) secretion and characerized by polyuria, is a common complication after neurosurgerical intervention and there is a lack of diagnostic criteria.Since the surgry casuses damage to patients' AVP-secreting neuronal cells, transient CDI (t-CDI) usually occurs 24-48h postoperatively and gradually resolves in about 10 days.However,permanent CDI (p-CDI) occurs in a small percentage of patients.Copeptin is a fragment of AVP, which has been shown to response the secretion of AVP.Multiple international studies have identified clinical applications for the use of copeptin to differentially diagnose adults with CDI , to assess electrolyte disturbances associated with AVP regulation, and to predict postoperative CDI after pituitary surgery.This study aims to investigate the trend of serum copeptin levels and its clinical value for postoperative CDI in pediatric patients after neurosurgerical intervention in ICU.

DETAILED DESCRIPTION:
In children and adolescents, the concentration distribution of copeptin has been gradually explored in recent years,but International studies have not yet shown the trend of copeptin levels in pediatric patients after neurosurgical intervention and its value in predicting CDI.

The primary objective of this study is to investigate the trend of serum copetin levels in ICU children after neurosurgerical intervention and compare differences of copeptide levels in children with CDI (t-CDI, p-CDI) and non-CDI. The secondary objective is to evaluate the optimal detection time and CUT OFF of copeptin in predicting the postoperative secondary CDI .

Blood sampling time points of serum copeptin levels are listed as follow:

presurgery(T0), 1h (T1), 1 day (T2), 2 days (T3), 3 days (T4), 4 days (T5), 5 day (T6) after surgury.

ELIGIBILITY:
Inclusion Criteria:

* Male and female,age ≥29 days and <18 years
* After neurosurgical intervention
* The patient agrees to comply with the requirements of the program, including follow-up visits and other related matters

Exclusion Criteria:

* Structural diseases of the genitourinary system (with the possibility of nephrogenic diabetes insipidus)
* Preoperative symptoms of diabetes insipidus
* Diabetes mellitus (HbA1c >8.5%)
* Drugs causing excessive drinking and urination (e.g., sodium-glucose cotransporter-2 inhibitors and diuretics)
* Lack of follow-up data after 3 months

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients after neurosurgical intervention in ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
C0-C6:The serum concentration of copeptin after NSI at T0 -T6 | Day0-6
  The serum concentration of copeptin after NSI at T0 -T6 to evaluate the trend of copetin level after NSI and its difference in children with CDI(t-CDI and p-CDI) and non-CDI

SECONDARY OUTCOMES:
ROC curve | Day0-6
  The curve of false positive rate and sensitivity with different critical point of serum copeptin level to diagnose CDI

CONTACTS AND LOCATIONS:
Overall Officials: guoping Lu, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China